CLINICAL TRIAL: NCT04881955
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [14C]-Ecopipam Following a Single Oral Capsule Dose in Healthy Male Subjects
Brief Title: Study of the Absorption, Metabolism, and Excretion of [14C]-Ecopipam in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emalex Biosciences Inc. (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EBS-101-HV-103
Record Dates: First submitted 2021-04-29; First posted 2021-05-11 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-Ecopipam (Experimental): Single oral capsule dose of 200 mg ecopipam HCl containing approximately 88.5 µCi of [14C]-ecopipam HCl
  Interventions: Drug: [14C]-Ecopipam

INTERVENTIONS:
Drug: [14C]-Ecopipam — [14C]-Ecopipam

SUMMARY:
Phase 1, single-center (United Kingdom), open-label, nonrandomized, single-dose study in healthy adult male subjects to assess the absorption, metabolism, and excretion of [14C]-Ecopipam in Healthy Male Subjects.

DETAILED DESCRIPTION:
This study will be a Phase 1, open-label, nonrandomized, single-dose study in healthy male subjects. Potential subjects will be screened to assess their eligibility to enter the study within 29 days prior to dose administration. Subjects will be admitted into the clinical research unit (CRU) on Day -1 and be confined to the CRU until at least Day 8 (Discharge). On Day 1, subjects will receive a single oral dose of 200 mg ecopipam HCl containing approximately 88.5 µCi of [14C]-ecopipam HCl. Subjects will be discharged when the following discharge criteria are met:

* plasma radioactivity levels below the limit of quantitation for 2 consecutive collections;
* ≥ 90% mass balance recovery; and
* ≤ 1% of the total radioactive dose is recovered in combined excreta (urine and feces) in 2 consecutive 24-hour periods in which collections occur. If discharge criteria are not met on Day 8, subjects will remain in the CRU and additional 24-hour collections (blood, urine, and feces) for total radioactivity will continue until these criteria are met, up to a maximum of Day 15.

ELIGIBILITY:
Inclusion Criteria:

* Males of any race between 35 and 55 years of age
* Body mass index between 18.0 and 30.0 kg/m2
* In good health
* Males will agree to use contraception
* Able to comprehend and sign an informed consent form
* History of a minimum of 1 bowel movement per day

Exclusion Criteria:

* History of significant medical illness
* History of clinically significant drug allergy
* History of a seizure disorder, not including infantile seizures
* History of stomach or intestinal surgery that would potentially alter absorption and/or excretion of orally administered drugs
* Clinically significant medical treatment within 8 weeks or infection treatment within 4 weeks of dosing
* Clinically significant ECG abnormality
* History of alcoholism or drug/chemical abuse within the previous 2 years or positive screening test
* Significant alcohol consumption
* Positive hepatitis panel and/or positive human immunodeficiency virus test
* Use of prohibited prescription, over-the-counter medications or natural health products
* Use of tobacco or nicotine-containing products within 3 months prior to Check-in or positive screening test
* Receipt of blood products within 2 months prior to Check in
* Recent donation of blood, plasma, or platelets prior to Screening
* Exposure to significant diagnostic, therapeutic or employment in a job requiring radiation exposure monitoring within 12 months prior to Check-in
* Evidence or history of active suicidal thoughts in the previous 5 years or have any lifetime history of a suicide attempt
* Not suitable for study in the opinion of the Principal Investigator

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Amount of radioactivity excreted in urine (Aeu) | Up to Day 15
  Up to 18 urine samples will be collected at the indicated time points
Cumulative radioactivity excreted in urine (Aeu) | Up to Day 15
  Up to 18 urine samples will be collected at the indicated time points
Amount of radioactivity excreted in feces (Aef) | Up to Day 15
  Up to 16 feces samples will be collected at the indicated time points
Cumulative radioactivity excreted in feces (Aef) | Up to Day 15
  Up to 16 feces samples will be collected at the indicated time points
Percentage of dose excreted in urine (feu) | Up to Day 15
  Up to 18 urine samples will be collected at the indicated time points
Percentage of dose excreted in feces (fef) | Up to Day 15
  Up to 16 feces samples will be collected at the indicated time points
Cumulative dose excreted in urine (feu) | Up to Day 15
  Up to 18 urine samples will be collected at the indicated time points
Cumulative dose excreted in feces (fef) | Up to Day 15
  Up to 16 feces samples will be collected at the indicated time points
Percentage of total radioactivity in total excreta (feces + urine) | Up to Day 15
  Up to 18 urine and feces samples will be collected at the indicated time points
Area under the plasma concentration versus time curve (AUC) from time zero extrapolated to infinity (AUC0-inf) | Up to Day 15
  Up to 28 blood samples will be collected at the indicated time points
AUC from time zero to the last quantifiable concentration (AUC0 last) | Up to Day 15
  Up to 28 blood samples will be collected at the indicated time points
Maximum observed concentration (Cmax) radioactivity feces + urine) | Up to Day 15
  Up to 28 blood samples will be collected at the indicated time points
Time of Cmax (Tmax) | Up to Day 15
  Up to 28 blood samples will be collected at the indicated time points
Apparent terminal elimination half-life (t1/2) | Up to Day 15
  Up to 28 blood samples will be collected at the indicated time points
Apparent total clearance (CL/F; ecopipam only) | Up to Day 15
  Up to 28 blood samples will be collected at the indicated time points
Apparent volume of distribution (Vz/F; ecopipam only) | Up to Day 15
  Up to 28 blood samples will be collected at the indicated time points
AUC0-inf of plasma ecopipam concentration relative to AUC0-inf of plasma total radioactivity (AUC0-inf Plasma ecopipam/Total Radioactivity Ratio) | Up to Day 15
  Up to 28 blood samples will be collected at the indicated time points
AUC0-inf of whole blood total radioactivity to AUC0-inf of plasma total radioactivity (AUC0 inf Blood/Plasma Ratio) | Up to Day 15
  Up to 28 blood samples will be collected at the indicated time points

SECONDARY OUTCOMES:
Percentage of ecopipam and metabolites to total radioactivity in plasma | Up to Day 15
  Up to 28 blood samples will be collected at the indicated time points
Percentage of ecopipam and metabolites to total radioactivity in urine and faeces | Up to Day 15
  Up to 18 urine and faeces samples will be collected at the indicated time points

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit Ltd., Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No